CLINICAL TRIAL: NCT03750760
Title: Early Alirocumab to Reduce LDL-C in Myocardial Infarction
Acronym: EARLY
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Changes in funding decision
Sponsor: Imperial College London (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18HH4627; 2018-002429-49 (Other Grant/Funding Number: R727-CV-17108)
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Infarction; Dyslipidemias
MeSH Terms: conditions — Myocardial Infarction; Dyslipidemias | interventions — alirocumab; Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alirocumab (enhanced care) (Active Comparator): Alirocumab (150 mg) administered by subcutaneous injection, every two weeks for 7 weeks.
  Atorvastatin (80 mg), oral administration daily.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin 80mg
- Atorvastatin (standard care) (Active Comparator): Atorvastatin (80 mg), oral administration daily. Ezetimibe (10 mg), oral administration daily, from week 4 if LDL-C is ≥ 70 mg/dL (1.8mmol/L) at week 4.
  Interventions: Drug: Atorvastatin 80mg; Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Alirocumab — PCSK9 (Proprotein Convertase Subtilisin Kexin Type 9) inhibitor antibody
  Other Names: Praluent
  Arms: Alirocumab (enhanced care)
Drug: Atorvastatin 80mg — 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statin)
Drug: Ezetimibe 10mg — Cholesterol absorption inhibitor
  Arms: Atorvastatin (standard care)

SUMMARY:
The EARLY trial is a phase IV, investigator initiated, international, multicentre study that will investigate if early use of alirocumab 150mg plus atorvastatin 80mg (enhanced care) will have a greater effect than atorvastatin 80mg (standard care) on the reduction of LDL-C at 2-weeks after a myocardial infarction (MI), in patients who start treatment within 24 hours of symptom onset.

A secondary goal is to assess the effects of enhanced care when compared to standard care which is either atorvastatin alone or atorvastatin plus ezetimibe, (the latter added at 4 weeks if LDL-C is ≥ 70mg/dL (1.8mmol/L), on the proportion of patients achieving an LDL-C goal of < 50mg/dL (1.29 mmol/L) at 7 weeks after an MI.

DETAILED DESCRIPTION:
Patients with Acute Coronary Syndrome (ACS), which includes myocardial infarction, are at high risk of recurrent ischaemic events (e.g. heart attacks), and death. The current standard treatment includes high dose statins to lower low-density lipoprotein cholesterol (LDL-C), also known as bad cholesterol, soon after admission. In some cases, following assessment after 1-3 months, administration of a second line cholesterol lowering therapy (ezetimibe) may be added if LDL-C levels remain high ≥ 70mg/dL (1.8mmol/L). Many guidelines advocate that following ACS high dose statins should be used as first line therapy. If LDL-C levels remain greater than 70mg/dL (1.8mmol/L) then additional add on therapy on statins could be considered for ACS patients.

Consented patients meeting the eligibility criteria for the EARLY trial will be randomised to enhanced care or standard care within 24hrs of symptom onset for MI. Patients randomised to enhanced care will receive alirocumab 150 mg on randomisation and then every 2 weeks during a 7-week treatment period. All patients will receive atorvastatin 80 mg. Patients randomised to standard care with an LDL-C level ≥ 70mg/dL (1.8mmol/L) at week 4 will receive ezetimibe 10 mg, in addition to atorvastatin 80 mg for the remaining duration of the treatment period.

All patients will be followed up for a two-week period after completing the 7-week treatment period (i.e. a total of 9 weeks to assess safety).

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or above
* Admitted to hospital for ST-Segment Elevation MI (STEMI) or non-ST-Segment Elevation MI (NSTEMI) (proven by electrocardiogram (ECG) or biomarker evidence of MI)
* Statin naïve prior to MI
* Local LDL-C measurement available within 24 hrs of chest pain with no more than 1 dose of statin
* Ability and willingness to give written informed consent and to comply with the requirements of the study

Exclusion Criteria:

* No ECG or biomarker evidence of MI
* Received more than one dose of statin during the index event prior to randomisation
* Contraindication to atorvastatin 80mg
* Contraindication to ezetimibe
* Contraindication to alirocumab
* Unwillingness or inability to comply with study requirements, particularly with respect to laboratory tests, specifically blood draws 24 and 48 hours after randomisation, and subsequent clinic visits
* New York Heart Association (NYHA) Class IV Heart Failure
* Unstable arrhythmia
* Subjects who in the opinion of investigator have a life expectancy of < 9 weeks
* Women of child bearing age who are not using at least 2 methods of contraception
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C in enhanced care group verses standard of care group at 2 weeks after randomisation | 2 weeks from baseline

SECONDARY OUTCOMES:
Percentage change in LDL-C at 7 weeks in enhanced care verses standard of care. | 7 weeks from baseline
Proportion of patients who achieve a LDL < 50mg/dL (1.29mmol/L) at week 2, 4 and 7 in enhanced care verses standard of care | 2, 4 and 7 weeks from baseline
Proportion of patients in standard of care who need ezetimibe 10 mg to be added in the standard of care pathway at week 4 | 4 weeks from baseline
Proportion of patients with reported adverse events (AEs) | 7 and 9 weeks from baseline
Proportion of patients with reported serious adverse events (SAEs) | 7 and 9 weeks from baseline
Proportion of patients with reported adverse events of special interest (AESIs) | 7 and 9 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Ray, Professor, Principal Investigator — Imperial College London
Locations (17):
- United Kingdom (17):
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - The Royal Bournemouth General Hospital, Bournemouth, Dorset
  - East Sussex Healthcare NHS Trust, Saint Leonards-on-Sea, East Sussex
  - Basildon Hospital, Basildon, Essex
  - St Mary's Hospital, London, Greater London
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Southampton General Hospital, Southampton, Hampshire
  - Northwick Park Hospital, Harrow, Middlesex
  - Hull Royal Infirmary, Hull, North Humberside
  - Queens Medical Centre, Nottingham, Nottinghamshire
  - St Peters Hospital, Chertsey, Surrey
  - East Surrey Hospital, Redhill, Surrey
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Queen Elizabeth Medical Centre, Birmingham, West Midlands
  - City Hospital, Birmingham, West Midlands
  - Worchestershire Royal Hospital, Worcester, Worcestershire
  - Northern General Hospital, Sheffield, Yorkshire

IPD SHARING:
Plan to Share IPD: No